CLINICAL TRIAL: NCT01182220
Title: Comparison of Ultrasound Guided L5/S1 Epidural Catheter Placement With Standard Epidural Catheter Placement: A Randomized Trial
Brief Title: Comparison of Ultrasound Guided Low Epidural Catheter Placement With Standard Epidural Catheter Placement
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-241-B
Record Dates: First submitted 2010-05-10; First posted 2010-08-16 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Labor Pain
Keywords: epidural; labor pain; ultrasound
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ultrasound L5/S1 catheter placement: Pt will have back scanned with Ultrasound and L5/S1 interspace localized for epidural placement.
- Control Group: Patients will have catheter placed after clinically evaluating the back as is done routinely resulting in mid lumbar catheter placement in general.

SUMMARY:
1. labor epidural quite often require bolus supplementation for better pain control control. Quite often this is due to sparing of sacral nerves.
2. If epidural is placed low in the L5/S1 interspace using ultrasound, this may minimize bolus requirement and improve patient labor experience.

DETAILED DESCRIPTION:
After consent patients will be randomized to one of the two groups: Control Group or the Experimental Group. Patients will be blinded to the group assignment.

In each subject prior to labor epidural placement, intravenous access will be obtained and if indicated fluid bolus will be given. There after heart and lung monitors will be placed. Procedure will be placed in sitting position. Standard epidural kit will be used.

In the Control Group the patient will be seated. Low back area will be prepped and draped in a sterile fashion. Lumbar interspaces will be identified clinically and epidural catheter will be inserted in the interspace deemed most appropriate. Epidural space will be accessed using loss of resistance to air technique. Once identified, a 20g open tip catheter will be placed can into the space.

In the Experimental Group, subjects back will be scanned with an Ultrasound probe. The interspace L5/S1, the lowest interspace in the spine will be identified and marked with the marker on the skin. Thereafter epidural catheter will be place using the exactly the same technique as used in the control group.

Once in place, catheter will be aspirated to rule out any intravascular placement. Thereafter a test dose composed of 45 mg lidocaine and 15 microgram epinephrine will be injected via the catheter to rule out any misplacement of catheter either in the intrathecal space or blood vessels. Once proper placement confirmed, catheter will be dose with 10 ml 0.25% bupivacaine in 5 ml boluses.

The extent of block before the surgery will be evaluated at 30 minutes post injection. Dermatomal level will be assessed on each side using ice. S1 and S2 dermatomal blockage will be specifically assessed on each side by testing lateral margin of each foot (S1 dermatome) and medial side of the popliteal fossa ( S2 dermatome).

Thereafter catheter will be connected to epidural solution containing 0.1% bupivacaine and 2 mic of Fentanyl per ml. Starting dose will be 10 ml per hr with bolus dose 5 ml q 30 minutes self administered by patient if needed.

If pain relief is inadequate top-up doses will be given consisting of 5 ml 0.25% bupivacaine times two 20 minutes part if needed. If no relief, dermatomal level will be reassessed. If ones sided or unequal, catheter will be pulled back I-2 cm and re-dosed with bupivacaine 0.25% 5 ml times two if needed over twenty minutes. If still no relief and inadequate level, catheter will be replaced.

Epidural catheter will be left in place till delivery. Patients will be clinically monitored as part of routine anesthetic management. Once they deliver catheter is removed by nurses in the labor and delivery unit and patients are sent to floor for recovery. Last evaluation will take place on post delivery day number one to evaluate patient satisfaction and address any concern patients may have.

Primary End points:

Primary purpose is to assess the ability of L5/S1 catheter to numb S1 or S2 dermatomes in comparison to routine placement of epidural catheter Secondary outcome to be assessed VAS, catheter manipulation or replacement between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Active labor age 18 or older

Exclusion Criteria:

* Known contraindications to epidural analgesia
* Any neurologic illness
* Fetal abnormalities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: active laboring patient without any complication requesting epdiural for pain control
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
1.Blocking of S1 and S2 dermatomes | 30 minutes after loading epidural
  After test dose and loading up of catheter, s1 and s2 dermatome blockage will be tested in L5/S1 epidural group vs conventionally placed epidural group. Idea is see if higher incidence of S1 and S2 blockage can be demonstrated in low epidural group.

SECONDARY OUTCOMES:
Number of top up doses for pain control throughout labor | from insertion till delivery average 8-24 hrs
  Better blocking of sacral dermatome should improve pain control and should result in clinically significant lower number of boluses.
Patient satisfaction | Evaluated on Post deliver day 1
  Improved pain control and less number of boluses should translate into better patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: TARIQ MALIK, MD, Principal Investigator — University of Chicago; Mohammed Minhaj, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States